CLINICAL TRIAL: NCT02038218
Title: A Phase II Trial: Safety and Tolerance of Intravenous 4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) in Patients With Malignancies Involving the Central Nervous System
Brief Title: Study of 4-Demethyl-4-cholesteryloxycarbonylpenclome (DM-CHOC-PEN) in Patients With Brain Tumors
Acronym: DM-CHOC-PEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DEKK-TEC, Inc. (Industry)
Collaborators: Tulane University (Other); Icahn School of Medicine at Mount Sinai (Other); Detroit Clinical Research Center (Other); National Cancer Institute (NCI) (NIH); Ochsner Health System (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTI-022; R44CA125871-03 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Primary Brain Tumors; Metastatic Malignant Neoplasm to Brain
Keywords: DM-CHOC-PEN; CNS; brain; melanoma; lung cancer; breast cancer; glioblastoma multiforme; primary brain tumors
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Lung Neoplasms; Breast Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DM-CHOC-PEN (Experimental): Two Cohorts of patients will be treated every once every 21 days with a single infusion of DM-CHOC-PEN as an out-patient. Patients will be divided into:
  Cohort 1: Patients with liver involvement or history of disease will be treated at a dose of 85.8 mg/m2 and;
  Cohort 2: Patients without liver involvement or history of liver disease, will be treated at a dose of 98.7 mg/m2.
  Patients in both cohorts will discontinue dosing with DM-CHOC-PEN when there are any unacceptable toxicities, progression of cancer or patient compliance.
  Interventions: Drug: 4-Demethyl-4-cholestryloxycarbonylpenclomedine

INTERVENTIONS:
Drug: 4-Demethyl-4-cholestryloxycarbonylpenclomedine — This will be an open-label, uncontrolled two-arm, multi-center study in patients with CNS involvement from melanoma, breast, lung cancers or primary malignancies of the CNS. Patients can be previously treated with radiation and systemic therapies and are eligible if they also have other sites of cancer involvement.
  Two Cohorts of patients will be treated every 21 days with a single infusion of DM-CHOC-PEN as an out-patient:
  Cohort 1: Patients with liver involvement or history of disease will be treated at a dose of 85.8 mg/m2 and;
  Cohort 2: Patients without liver involvement or history of liver disease, will be treated at a dose of 98.7 mg/m2.
  Patients in both cohorts will discontinue dosing with DM-CHOC-PEN when there are any unacceptable toxicities, progression of cancer or patient compliance.
  Other Names: DM-CHOC-PEN

SUMMARY:
DM-CHOC-PEN is a polychlorinated pyridine cholesteryl carbonate that has demonstrated antineoplastic activities in patients with advanced cancers - melanoma, lung, breast and glioblastoma multiforme (GBM) involving the CNS during a Phase I study. These findings support the preclinical responses seen in mice bearing intracerebrally implanted human breast and GBM tumor xenografts. Toxicity was acceptable - hyperbilirubinemia (in patients with liver disease and/or liver metastasis). No hematological, renal, cardiovascular, behavioral or cognitive impairment/neurotoxicities were noted during the Phase I human trial or in previous pre-clinical studies.

The drug is available for use as a soy bean oil/egg yolk lecithin/glycerin water emulsion; the latter continues to be chemically and biologically stable and safe.

Patients with advanced lung, breast and melanoma cancers spread to the CNS and primary CNS malignancies will be eligible for enrollment and treatment, providing the required blood and other eligibility requirements are met. The trial will be 2-tiered - patients with liver involvement vs. non-liver involvement will be treated with different doses of the drug.

The trial is open and patients are currently being enrolled and treated with the protocol.

DETAILED DESCRIPTION:
DM-CHOC-PEN has been selected for Phase II intravenous studies in the treatment of patients with advanced malignancies with central nervous system measurable disease based on the improved PFS and objective responses seen for patients treated during the Phase I DTI-021 trial and the manageable toxicities noted. Melanoma, breast and lung cancers involving the CNS have responded to DM-CHOC-PEN in the Phase I study, thus the basis for the choice of tumors to be treated in the Phase II trial. Currently, the opinion is that the drug is penetrating the blood brain barrier (BBB) attached to rbcs and released intracerebrally in tumor masses in situ.

The trial will be carefully monitored, and if a cancer type has >3 confirmed responders in the first 18 evaluable patients (Stage -1 enrollment); accrual will be expanded for that tumor type with a goal of 7/43 for achieving an 80% power at the 5% level of significance (Stage-2 enrollment) with unacceptable response rate (P0) 0.1 and desirable response rate (P1) 0.25. Thus, each arm will have a 2-stage design. This will allow resources to be directed to the most promising areas - selection of 1 or 2 tumor types to develop via additional trial studies. A desirable response rate is 25% or better. The above is for each tumor type - lung, breast, melanoma and GBM.

In summary, for any tumor type or treatment sub-group, a response rate of <15% or a rate of "possibly treatment-related Gr-3/4 toxicities" of >25% will be considered unacceptable and enrollment in the respective tumor type category will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological proof of a cancer - melanoma, breast, or lung cancer - which has spread to the CNS or glioblastoma (GBM) or other primary malignant neoplasm of the CNS which has been treated with standard treatments, which may include radiation, and must be measurable (RECIST).
* Patients must have life expectancy of at least 12 weeks and a Karnofsky performance score: > 60 % (or a Zubrod performance status of < 2).
* The age limit - 18 or older. Gender is not a criterion.
* All patients must be off previous chemo- and/or radiotherapy for at least three (3) weeks prior to entrance into the study and have recovered from any toxic effects induced by such treatment(s); no nitrosourea type drug or ipilumimab treatments are permitted within the last six (6) weeks prior to enrollment. No major surgery within 14 days of enrollment. Patients may continue to receive anti-estrogen/steroid therapy that has been initiated at least eight weeks prior to enrollment in the study.
* Patients should have adequate bone marrow function defined as a peripheral WBC >3,000/mm3 with an ANC >1500/mm3 and a platelet count >100,000/mm3.
* Patients should have hepatic function (alkaline phosphatase, AST and ALT) < ULN and renal functions with serum creatinine - <1.5 x UNL. If a patient has liver metastasis and/or a history of liver disease - they will receive a lower dose of the drug per treatment protocol.
* Patients should not be allergic to eggs or soy beans. Patients must be medically, psychologically and neurologically stable and have triplicate baseline ECG's with a mean QTc interval <500 ms and >300 ms and neither a history of congenital prolonged or short QT syndrome. Patients with a history of cardiac disease must be stable.
* Patients must understand the nature of the study and be willing to sign an informed consent that complies with the investigator/DEKK-TEC policies and approved by the Human Investigation Review Committee. Patients must have CNS involvement - from a malignancy. Lung cancer may be either small cell or non-small cell.

Exclusion Criteria:

* Patients with concurrent severe and/or uncontrolled medical co-morbidities - including active infections, unstable uncontrolled diabetes, cardiovascular and pulmonary, renal, psychiatric or social conditions that could compromise the safety or compliance of treatment are not eligible.
* Concomitant chemotherapy or radiotherapy is not permitted.
* Pregnant or lactating females are excluded. Women of childbearing age, and their sexual partners, must use an effective contraception program. Males who are having sexual relations with women capable of child bearing must use the barrier birth control while on the study and for 3- months after the last dose of the study drug.
* Patients taking CYP3A4 inducers or inhibitors are not eligible since it is not known whether the study drug is metabolized through this pathway. The following CYP3A4 inhibitors/inducers are not permitted during the trial - the azole antifungal - fluconazole, erythromycin, phenobarbital, verapamil.
* Patients taking the following medications may experience QT/QTc interval prolongation and are not eligible for the trial - most anti-arrhythmia drugs (incl. amiodarone), erythromycin, quinolone antibiotics, ketoconazole, Zithromax, and phenothiazine and will be denied enrollment in the study. The possible interactions of these drugs and DM-CHOC-PEN have not been established. Patients receiving these drug will only be eligible if they discontinue the drugs and have an acceptable ECG.
* Coagulopathies - patients requiring full dose anticoagulation with warfarin are excluded, however, patients stable and on other anticoagulants can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee R Morgan, MD, PhD, Study Director — DEKK-TEC, Inc.
Locations (3):
- United States (3):
  - Tulane University Medical Center, New Orleans, Louisiana
  - Detroit Clinical Research Centers, Lansing, Michigan
  - The University of Texas Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
As approved by the NCI
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Five years
Access Criteria: Per contact with the Study Director
URL: https://dekk-tec.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study completed - Tulane Medical Center (2017-19), Detroit Research Center (Lansing, Detroit and Owasso) 2017-19, Mt Sinai Medical Center, NYNY, 2014-18 and Ochsner Medical Centers (New Orleans, 2017-19.
Pre-assignment Details: Patients with cancer involving the CNS were treated with intravenous DM-CHOC-PEN. The drug is metabolized by the liver. Abnormal neurological and hepatic values excluded the patients from treatments. If the patients were on steroids, this also excluded treatments. Steroids initiate the break down of DM-CHOC-PEN.
Groups:
- DM-CHOC-PEN - Arm 1: Cohort 1: Patients without liver involvement or history of liver disease, will be treated at a dose of 98.7 mg/m2.
  Patients in both Arms 1 & 2 will discontinue dosing with DM-CHOC-PEN when there are any unacceptable toxicities, progression of cancer or patient compliance.
  4-Demethyl-4-cholestryloxycarbonylpenclomedine: This will be an open-label, uncontrolled two-arm, multi-center study in patients with CNS involvement from melanoma, breast, lung cancers or primary malignancies of the CNS. Patients can be previously treated with radiation and systemic therapies and are eligible if they also have other sites of cancer involvement.
  Two Cohorts of patients will be treated every 21 days with a single infusion of
- DM-CHOC-PEN - Arm 2: Cohort 2: Patients with liver involvement or history of disease will be treated at a dose of 85.8 mg/m2; 5 patients were in this group
Period: Overall Study
Arm/Group | DM-CHOC-PEN - Arm 1 | DM-CHOC-PEN - Arm 2
Started (The aim of the project was that the drug was acceptable in patients with liver disease.) | 22 (Drug tolerated - Arm 1: No liver disease - 98.7 mg/m2. No alterations of liver functions.) | 7 (Drug tolerated - Arm 2: liver involvement - 85.5 mg/m2. No alterations of liver functions.)
Completed (22 patients were treated) | 22 (22 patients are included in a publication in progress) | 7 (5 patients are included in a publication in progress)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with liver complications lower dose
Groups:
- ARM 1: Arm-1: Patients with without liver involvement or history of liver disease, will be treated at a dose of 98.7 mg/m2.
  Patients will be treated every once every 21 days with a single infusion of DM-CHOC-PEN as an out-patient.
  4-Demethyl-4-cholestryloxycarbonylpenclomedine: This will be an open-label, uncontrolled two-arm, multi-center study in patients with CNS involvement from melanoma, breast, lung cancers or primary malignancies of the CNS.
- ARM 2: Arm-2: Patients with liver involvement or history of liver disease, will be treated at a dose of 85.8mg/m2.
  Patients will be treated every once every 21 days with a single infusion of DM-CHOC-PEN as an out-patient.
  4-Demethyl-4-cholestryloxycarbonylpenclomedine: This will be an open-label, uncontrolled two-arm, multi-center study in patients with CNS involvement from melanoma, breast, lung cancers or primary malignancies of the CNS.
- Total: Total of all reporting groups
Arm/Group | ARM 1 | ARM 2 | Total
Number analyzed (Participants) | 22 | 7 | 29
Age, Categorical [Count of Participants; unit: Participants] — 18 years of age and greater
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 22 | 6 | 28
    >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (8) | 61 (10) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 14 | 5 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 7 | 29
Average Initial Tumor Diameter [Mean (Standard Deviation); unit: cm] | 2.8 (1.3) | 2.6 (0.8) | 2.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Diameter
Description: Tumor Diameter from patient scans
Time Frame: Until remission or off treatment due to progression
Population: Mean Tumor size after Treatment
Measure: Mean (Standard Deviation); unit: cm
Groups:
- DM-CHOC-PEN - Arm 1: Cohort 1: Patients without liver involvement or history of liver disease, will be treated at a dose of 98.7 mg/m2.
  Patients will discontinue dosing with DM-CHOC-PEN when there are any unacceptable toxicities, progression of cancer or patient compliance.
  4-Demethyl-4-cholestryloxycarbonylpenclomedine: This will be an open-label, uncontrolled two-arm, multi-center study in patients with CNS involvement from melanoma, breast, lung cancers or primary malignancies of the CNS. Patients can be previously treated with radiation and systemic therapies and are eligible if they also have other sites of cancer involvement.
- DM-CHOC-PEN - Arm 2: Cohort 2: Patients with liver involvement or history of disease will be treated at a dose of 85.8 mg/m2.
  Patients will discontinue dosing with DM-CHOC-PEN when there are any unacceptable toxicities, progression of cancer or patient compliance.
  4-Demethyl-4-cholestryloxycarbonylpenclomedine: This will be an open-label, uncontrolled multi-center study in patients with CNS involvement from melanoma, breast, lung cancers or primary malignancies of the CNS. Patients can be previously treated with radiation and systemic therapies and are eligible if they also have other sites of cancer involvement.
Arm/Group | DM-CHOC-PEN - Arm 1 | DM-CHOC-PEN - Arm 2
Number analyzed (Participants) | 22 | 7
cm | 2.7 (1.1) | 4.4 (0.8)

2. Primary Outcome: Overall Survival
Description: Overall survival in months
Time Frame: Until death
Measure: Median (Standard Deviation); unit: Months
Arm/Group | DM-CHOC-PEN - Arm 1 | DM-CHOC-PEN - Arm 2
Number analyzed (Participants) | 22 | 7
Months | 11 (8) | 8 (3)

ADVERSE EVENTS:
Time Frame: Data was collected over 2.5 years
Groups:
- ARM 1: Patients without liver involvement
- ARM 2: Patients with liver involvement
Arm/Group | ARM 1 | ARM 2
All-Cause Mortality (participants affected / at risk) | 19/22 | 7/7
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/7
Other Adverse Events (participants affected / at risk) | 3/22 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 (N=22) | ARM 2 (N=7)
Headache (Nervous system disorders) | 1 (1) | 0
Seizures (Nervous system disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The study was to evaluate the effects of DM-CHOC-PEN on brain tumor lesions. All patients had cancer involving the central or spinal NS; NSCLC responded best. However, most patients had cancer out side of the brain, which was the cause of death.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes